CLINICAL TRIAL: NCT06370104
Title: Treating Suicidality Remotely: a Randomized Controlled Trial of Brief Cognitive Behavioral Therapy for Suicide Prevention Delivered Via Chat or Phone
Brief Title: Treating Suicidality Remotely
Acronym: TREASURE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 113 Suicide Prevention (Other)
Collaborators: Amsterdam UMC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL85041.018.23
Record Dates: First submitted 2024-04-08; First posted 2024-04-17 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Suicide Attempt
Keywords: suicide; attempts; ideation; telehealth; e-health; remote; cbt; self-help
MeSH Terms: conditions — Suicide, Attempted; Suicide; Color Vision Defects

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trial with a 1:1 allocation ratio.
Who Masked: Outcomes Assessor
Masking Description: Participants are not blind to the treatment condition, but are unaware which is the experimental condition and which the control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Brief Cognitive Behavioral Therapy for Suicide Prevention (Experimental): Participants in the experimental condition will be treated with online CBT-SP, a personalized intervention of approximately 12 sessions via chat or phone, in which therapist and client create a safety plan, try to restrict the access to lethal means and use a narrative assessment of a recent suicidal crisis to create a case formulation. This case formulation is then used to choose from several treatment modules, such as dealing with unhelpful thoughts and reducing sleep problems.
  Interventions: Behavioral: Brief Cognitive Behavioral Therapy for Suicide Prevention
- Remote Semi-guided self-help course (Active Comparator): Participants in the control group will be treated with a self-help course, in which they are given psychoeducation on suicidal thoughts, create a safety plan and are thought several techniques from cognitive therapy, such as cognitive restructuring and worry times. The course consists of 6 sessions, on which subjects receive feedback from a therapist. In this study, feedback will be given in a live conversation with the therapist via chat or phone, instead of via e-mail, to increase safety and reduce the difference in attention between the groups.
  Interventions: Behavioral: Living under control

INTERVENTIONS:
Behavioral: Brief Cognitive Behavioral Therapy for Suicide Prevention — see arm description
  Arms: Remote Brief Cognitive Behavioral Therapy for Suicide Prevention
Behavioral: Living under control — see arm description
  Other Names: Living with deadly thoughts
  Arms: Remote Semi-guided self-help course

SUMMARY:
Background: Practical and psychological barriers make it difficult for people with Suicidal Thoughts and Behaviors (STBs) to get professional help. Online interventions have the potential to overcome many of these barriers, but the online interventions to date have produced small or short-lived effects and have only been found to reduce suicidal thoughts, not behaviors. This is a crucial limitation, since previous studies have shown that interventions that reduce suicidal thoughts often do not prevent suicide attempts, and vice versa.

Methods: A fully remote randomized controlled trial will be conducted in which 364 participants of 16 years and older will be recruited through the website of a suicide prevention helpline in the Netherlands and randomized with an allocation ratio of 1:1 to either Brief Cognitive Behavioral Therapy for Suicide Prevention (BCBT-SP) or a semi-guided online self-help course that has previously been found superior to waitlist in reducing suicidal thoughts. The primary outcome of the study is the number of suicide attempts, measured with the Columbia Suicide Severity Rating Scale. Secondary outcomes are self-reported suicidal ideation, healthcare utilization, treatment satisfaction, adverse effects, and quality of life. All outcomes will be assessed at baseline, immediately after the treatment and at 18 months follow-up.

Discussion: If remote BCBT-SP proves effective, the findings of this study will add to the evidence base of BCBT-SP as one of very few psychological interventions with replicated effectiveness in preventing suicide attempts and provide the first evidence to date that remote interventions cannot only reduce suicidal thoughts, but also prevent suicidal behavior.

ELIGIBILITY:
Inclusion Criteria:

* 16 years or older
* Currently living in The Netherlands
* Any type of STBs in the past 4 weeks

Exclusion Criteria:

* Insufficient mastery of the Dutch language
* Previously engaged in 113 Suicide Prevention's Online Therapy or Self-help course
* Currently seeing a mental health professional at least once every 3 weeks, other then a general practitioner or general practice based nurse practitioner ('POH-GGZ')
* Not able to engage in online therapy, for instance because of severe mood disorders or psychotic symptoms, based on the clinical impression of the research assistant and a supervisor

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2028-04-25 (Estimated); Study Completion 2028-04-25 (Estimated)

PRIMARY OUTCOMES:
Number of suicide attempts | 18-months follow-up
  Number of fatal and non-fatal suicide attempts, identified through the Columbia Suicide Severity Rating Scale (C-SSRS; non-fatal attempts), a contact provided by the participant or Statistics Netherlands (fatal attempts).

SECONDARY OUTCOMES:
Severity of suicidal ideation | 18-months follow-up
  Severity of suicidal ideation as measured with the suicidal ideation subscale of the Suicide Severity Rating Scale. This sub scale results in a score from 1-5 based on the most severe type of suicidal ideation endorsed by the subject. For this study, subjects who do not report any suicidal ideation are assigned a score of 0.
Severity of suicidal Thoughts and Behaviors Composite | 18-months follow-up
  A total score for STB severity will be derived from the Columbia Suicide Severity Rating Scale: subjects who report no suicidal thoughts or behaviors will be assigned a score of 0; subjects who report suicidal thoughts but not behaviors a score of 1-5, depending on their rating on the suicidal ideation subscale described above; subjects who report preparatory behavior but no attempt a score of 6; subjects who report an aborted attempt a score of 7; subjects who report an interrupted attempt a score of 8; and subjects who report a non-lethal attempt a score of 9. Subjects who have made a lethal attempt will be assigned a score of 10.
Treatment satisfaction | post-treatment (approximately 12 weeks after the start of treatment)
  Treatment satisfaction as measured with the Client Satisfaction Questionnaire 8 (CSQ-8). The subject's scores on the 8 items of the scale are summed up, resulting in a score between 8 and 32, with higher values indicating higher satisfaction.
Adverse effects | post-treatment (approximately 12 weeks after the start of treatment)
  Adverse effects as measured with the 20-item version of the Negative Effects Questionnaire (NEQ). The mean number of negative effects that clients report and attribute to the treatment is calculated.
Co-occuring mental health issues | 18-months follow-up
  Co-occuring mental health issues as measured with the MINI neuropsychiatric interview - simplified. Two scores are calculated:
  * the mean number of symptoms per client
  * the mean number of classifications per client
Quality of life | 18-months follow-up
  Quality of life as measured with the Mental Health Quality of Life Questionnaire. An overall index score is calculated by summing the scores of the seven questions. This index score can vary from 0 to 21, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- 113 Suicide Prevention, Amsterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: within two years after data collection has been completed